CLINICAL TRIAL: NCT06386133
Title: Chronic Fatigue in Multiple Sclerosis: Validating Clinical Performance, Economic, and Organizational Benefits of MSCopilot Boost Compared to Standard Care
Brief Title: Chronic Fatigue in Multiple Sclerosis: MS Copilot Boost Solution Compared to Standard Care
Acronym: MSBoost
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ad scientiam (Other)
Collaborators: URC-ECO Clinical trial unit on health Economics, Hotel-Dieu Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MS Boost
Record Dates: First submitted 2024-04-16; First posted 2024-04-26 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2024-10

CONDITIONS: Multiple Sclerosis; Fatigue Syndrome, Chronic
Keywords: Mobile application; Digital monitoring; Fatigue management; Multiple sclerosis
MeSH Terms: conditions — Multiple Sclerosis; Fatigue Syndrome, Chronic | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Boost group: Use of MSCopilot Boost and wear of an actimeter during the whole study participation duration.
  Control group: Standard practice and wear of an actimeter during the whole study participation duration.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Boost Group (Experimental): The Boost Group will have the MSCopilot Boost mobile application and follow personalized fatigue management advices and physical activity program
  Interventions: Device: MS Boost
- Control Group (Active Comparator): The Control Group will follow standard of care with general fatigue advices
  Interventions: Other: Standard of care

INTERVENTIONS:
Device: MS Boost — remote monitoring digital tool based on functional tests (walking, dexterity, vision and cognition). These digital tests may be combined with a fatigue assessment via questionnaires and, if needed, a telerehabilitation program. This program includes an algorithm comprising fatigue management advice and/or physical activity recommendations personalised to the patients, aimed at improving fatigue-related symptoms. The patient can use the telerehabilitation program without supervision
  Arms: Boost Group
Other: Standard of care — General fatigue tips are given to patients who suffering from chronic fatigue such as stop smoking, eat a healthy diet...
  Arms: Control Group

SUMMARY:
The main objective of the MS Boost study is to demonstrate the superiority of MSCopilot Boost over standard practice in reducing the impact of fatigue on Patients with Multiple Sclerosis (MS).

The secondary objectives include validating MSCopilot Boost clinical performance in reducing fatigue and its impact as well as evaluating its functional tests performance and its safety of use. The investigation team will also investigate the effects of MSCopilot Boost on patient symptoms, functional parameters and physical activity levels. The investigation team will evaluate patients and healthcare professionals' perceived clinical benefit as well as adherence, satisfaction and user experience related to the mobile application and the web portal. Ultimately, the investigation team will define the medico-economic and organizational impact of the MSCopilot Boost solution.

Patients' expected benefits are the access to additional clinical tests not routinely performed, covering dimensions not addressed by standard tests like the EDSS for example; a remote monitoring of functional tests similar to those of the modified MSFC with the possibility of adding an evaluation of fatigue through digital questionnaires; improvement of symptoms related to MS fatigue through access to a personalised tele-rehabilitation program.

Healthcare professionals' expected benefits are to track objective measures of key functional symptoms of the disease between consultations, supporting MS patients' management and to gain time by providing a "big picture" of the patient's condition over time.

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is an autoimmune, inflammatory disease of the central nervous system that causes unpredictable neurological symptoms. It is the leading cause of non-traumatic disability in young adults in France. MS often leads to mobility impairments, visual problems (26% of patients), cognitive dysfunction (40-70%) and chronic fatigue, which affects more than 70% of patients. Fatigue, a major problem for 55% of patients, reduces energy, affects work capacity and increases sickness absence. Despite its importance, common clinical tools such as the EDSS and MSFC-4 do not assess fatigue.

MS-related fatigue is multifactorial, influenced by disease phenotype, comorbidities (e.g. depression, pain, sleep problems) and lifestyle factors. Fatigue assessments such as the Fatigue Severity Scale (FSS) and the Modified Fatigue Impact Scale (MFIS) are commonly used, but have validity issues and often require additional qualitative methods.

There is no clear consensus on the management of fatigue in MS. Pharmacological treatments show inconsistent results and non-pharmacological methods, particularly physical activity, are promising. Moderate exercise and resistance training improve symptoms and fitness, but no single exercise regimen is superior, so individualised approaches are needed. Multidisciplinary management combining physical activity, behavioural therapies and sometimes medications is increasingly recommended.

Most people with MS do not meet physical activity guidelines, highlighting the need for tailored exercise programmes. Mobile applications for remote monitoring and self-management offer promising solutions to enable patients to maintain activity and manage symptoms between medical visits.

Ad Scientiam has developed MSCopilot Boost, a medical software device that supports remote monitoring and management of MS symptoms. It includes a smartphone app with functional tests for walking, dexterity, vision, cognition and fatigue, and a telerehabilitation programme with personalised advice. Healthcare professionals can track patient progress via a web portal, making MSCopilot Boost a complementary tool to support consultations, rather than a stand-alone diagnostic device.

The primary objective of the MS Boost study is to demonstrate the efficacy of MSCopilot Boost in reducing the impact of fatigue in people with MS. Secondary objectives include evaluating its performance in reducing fatigue, improving functional testing, ensuring safety, and assessing its impact on symptoms and physical activity levels. The study also aims to measure patient and healthcare professional satisfaction, adherence and user experience with the app and web portal, and to define its organisational and economic impact.

Patients could benefit from additional clinical tests, real-time monitoring of functional parameters and a personalised fatigue management programme, while healthcare professionals would gain insight into patients' conditions over time, enabling more efficient management of MS-related symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Aged over 18 years
* With a confirmed MS diagnosis according to 2017 McDonald's revised criteria
* Having an EDSS score comprised between 0 and 6.5
* With a fatigue score ≥ 43 on MFIS scale
* Able to walk with or with walking aids
* Owning a personal smartphone with a mobile operating system version higher than 14 for IOS (iPhone) and 8 for Android
* Able to read the language in which the mobile application is available and able to understand pictograms
* Affiliated to a social security system
* Having signed the free and informed consent
* Having accepted to wear an actimeter during the whole duration of study participation
* Having been on a stable disease-modifying therapy for MS for at least 6 months.

Exclusion Criteria:

* Psychiatric disorder, major visual or cognitive deficiency, as assessed by the investigator
* Participation in an exercise reconditioning program at a rehabilitation center within the 6 weeks prior to inclusion
* Major comorbidities that could influence fatigue management (lupus, rheumatoid arthritis, chronic obstructive pulmonary disease, chronic fatigue syndrome, etc).
* Contraindication to physical activity:
* History of cardiac events:
* Abnormal cardiac examination at last medical check-up.
* Palpitations, tachycardia or irregular heartbeat
* Pain and shortness of breath:
* Cramp-like pain in the lower limbs when walking, disappearing when walking stops, except for MS-related pain (neuropathic or spastic).
* Chest pain
* Shortness of breath at rest (appearing or worsening in the lying position)
* Shortness of breath during low-intensity exercise or usual activities
* Pain, discomfort or heaviness in the chest at rest or during exertion
* Unstable chronic diseases :
* Unstable metabolic disease
* Unstable renal disease
* Uncontrolled chronic disease
* Ankle edema
* Dizziness or syncope
* Having received fampridine, corticosteroid therapy or therapeutic cannabis within the 2 months prior to inclusion.
* Psychoactive substances and/or alcohol consumption likely to influence test performance (investigator's judgment).
* Patients confined to bed or whose daily activity is less than 2 hours.
* Persons under guardianship or curatorship.
* Pregnant or breast-feeding women.
* Subjects who have participated in another clinical study within 30 days prior to selection, or who are participating in another study that, in the opinion of the investigator, could interfere with full participation in the study or confound the participant's assessment or the study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Estimated)
Dates: Start 2026-12-01 (Estimated); Primary Completion 2027-08-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
To demonstrate that MSCopilot Boost is superior to standard practice in reducing the impact of fatigue on Patients with Multiple Sclerosis | During the first in-clinic visit (Day 0) and the end of study visit in-clinic (Day 270)
  Comparison of mean decrease in the Modified Fatigue Impact Scale score (MFIS) between Boost and Control groups from Day 0 to Day 270 .
  The criteria will be considered as positive if the Boost group shows a mean decrease of at least a 7 point in Day 270 score, compared to the Control group.
  The score ranges from 0 to 84, with a higher score indicating a worse outcome.

SECONDARY OUTCOMES:
To evaluate the impact of fatigue in both groups. | During the first in-clinic visit (Day 0), during the in-clinic follow-up visits (Day 90 and Day180) and the end of study visit in-clinic (Day 270)
  Measure of the mean decrease in Modified Fatigue Impact Scale score:
  * In the Boost group
  * Between Day 0 and Day 90
  * Between Day 0 and Day 180
  * Between Day 0 and Day 270
  * In the Control group
  * Between Day 0 and Day 90
  * Between Day 0 and Day180
  * Between Day 0 and Day 270
  The score ranges from 0 to 84, with a higher score indicating a worse outcome.
To compare the effect of MSCopilot Boost in reducing fatigue impact compared to standard practice (Short term and Medium term) | During the first in-clinic visit (Day 0) and during the in-clinic follow-up visits (Day 90 and Day180)
  Comparison of the mean decrease in Modified Fatigue Impact Scale score:
  * Between Day 0 and Day 90
  * Between Day 0 and Day 180
  The score ranges from 0 to 84, with a higher score indicating a worse outcome.
To compare the fatigue impact between the two groups. | During the in-clinic follow-up visits (Day 90 and Day180) and the end of study visit in-clinic (Day 270)
  Comparison of Modified Fatigue Impact Scale score between the two groups:
  * At Day 90
  * At Day 180
  * At Day 270
  The score ranges from 0 to 84, with a higher score indicating a worse outcome.
To compare the effect of MSCopilot Boost in reducing perceived fatigue compared to standard practice. | During the first in-clinic visit (Day 0), during the in-clinic follow-up visits (Day 90 and Day180) and the end of study visit in-clinic (Day 270)
  Comparison of the mean fatigue score by using a visual analog scale (from daily activities impact questionnaire) between the two groups:
  * Between Day 0 and Day 90
  * Between Day 0 and Day 180
  * Between Day 0 and Day 270
  Score ranges from 0 (not impacted) to 10 (very impacted), with a higher score indicating a worse outcome.
Correlation of MSCopilot Boost functional test performed autonomously at home with its standard counterpart performed under supervised conditions at the hospital. | During the first in-clinic visit (Day 0) and the first at-home visit (Day 1)
  Pearson correlation coefficient to evaluate the correlation between the active Mobile Walking Perimeter Test (in meter) performed at Day 1 (at home) with the standard test Timed 25 Foot Walk (in seconds) performed at Day 0 (at the hospital) in the Boost group.
Correlation of MSCopilot Boost functional test performed autonomously at home with its standard counterparts performed under supervised conditions at the hospital. | During the first in-clinic visit (Day 0) and the first at-home visit (Day 1)
  Pearson correlation coefficient to evaluate the correlation between the active Mobile Walking Endurance Test (in meters) performed at Day 1 (at home) with the standard test Timed 25 Foot Walk (in seconds) performed at Day 0 (at the hospital) in the Boost group.
Correlation of MSCopilot Boost functional test performed autonomously at home with its standard counterpart performed under supervised conditions at the hospital. | During the first in-clinic visit (Day 0) and the first at-home visit (Day 1)
  Pearson correlation coefficient to evaluate the correlation between the active Mobile Dexterity Test (in seconds) performed at Day 1 (at home) with the standard test 9 Hole Peg Test (in seconds) performed at Day 0 (at the hospital) in the Boost group.
Correlation of MSCopilot Boost functional test performed autonomously at home with its standard counterpart performed under supervised conditions at the hospital. | During the first in-clinic visit (Day 0) and the first at-home visit (Day 1)
  Pearson correlation coefficient to evaluate the correlation between the active Mobile Cognition Test (score) performed at Day 1 (at home) with the standard Symbol Digit Modalities Test (score) performed at Day 0 (at the hospital) in the Boost group.
Correlation of MSCopilot Boost functional test performed autonomously at home with its standard counterpart performed under supervised conditions at the hospital. | During the first in-clinic visit (Day 0) and the first at-home visit (Day 1)
  Pearson correlation coefficient to evaluate the correlation between the active Mobile Vision Test (number stated) performed at Day 1 (at home) with the standard Sloan Low Contrast Letter Acuity Test (number of letter stated) performed at Day 0 (at the hospital) in the Boost group.
  Higher is the number of letter or number stated, better is the outcome.
Correlation of the answers of MSCopilot Boost questionnaire performed autonomously with its standard counterpart performed under supervised conditions at the hospital | During the first in-clinic visit (Day 0) and the end of study visit in-clinic (Day 270)
  Intra class correlation coefficient (ICC) to assess the correlation between electronic and standard version of the Daily activities impact questionnaire completed by patients at Day 0 and Day 270.
  The score ranges from 0 to 10, with higher score meaning worse outcome.
Correlation of the answers of MSCopilot Boost questionnaire performed autonomously with its standard counterpart performed under supervised conditions at the hospital | During the first in-clinic visit (Day 0) and the end of study visit in-clinic (Day 270)
  Intra class correlation coefficient (ICC) to assess the correlation between electronic and standard version of the Modified Fatigue Impact Scale-5 questionnaire completed by patients at Day 0 and Day 270.
  Score ranges from 0 to 20, with higher score meaning worse outcome.
Correlation of the answers of MSCopilot Boost questionnaire performed autonomously with its standard counterpart performed under supervised conditions at the hospital | During the first in-clinic visit (Day 0) and the end of study visit in-clinic (Day 270)
  Intra class correlation coefficient (ICC) to assess the correlation between electronic and standard version of the Sleep questionnaire completed by patients at Day 0 and Day 270.
Correlation of the answers of MSCopilot Boost questionnaire performed autonomously with its standard counterpart performed under supervised conditions at the hospital | During the first in-clinic visit (Day 0) and the end of study visit in-clinic (Day 270)
  Intra class correlation coefficient (ICC) to assess the correlation between electronic and standard version of the Mental well-being (PHQ-4) questionnaire completed by patients at Day 0 and Day 270.
  Score ranges from 0 to 12, with higher score meaning worse outcome.
Correlation of the answers of MSCopilot Boost questionnaire performed autonomously with its standard counterpart performed under supervised conditions at the hospital | During the first in-clinic visit (Day 0) and the end of study visit in-clinic (Day 270)
  Intra class correlation coefficient (ICC) to assess the correlation between electronic and standard version of the Physical Activity Level questionnaire (IPAQ) completed by patients at Day 0 and Day 270.
Correlation of the reproductibility of MSCopilot Boost functional test from the hospital to home. | During the first in-clinic visit (Day 0), the first at-home visit (Day 1), the follow-up visit at-home (Day 89) and the follow-up visit in-clinic (Day 90)
  Intraclass correlation coefficient (ICC) to assess the reproducibility between the Mobile Walking Perimeter Test (in meters) performed at hospital and at home
  * At Day 0 and Day 1
  * At Day 89 and Day 90
  Higher is the distance, better is the outcome.
Correlation of the reproductibility of MSCopilot Boost functional test from the hospital to home. | During the first in-clinic visit (Day 0), the first at-home visit (Day 1), the follow-up visit at-home (Day 89) and the follow-up visit in-clinic (Day 90)
  Intraclass correlation coefficient (ICC) to assess the reproducibility between the Mobile Dexterity Test (in seconds) performed at hospital and at home
  * At Day 0 and Day 1
  * At Day 89 and Day 90
  Shorter is the time, better is the outcome.
Correlation of the reproductibility of MSCopilot Boost functional test from the hospital to home. | During the first in-clinic visit (Day 0), the first at-home visit (Day 1), the follow-up visit at-home (Day 89) and the follow-up visit in-clinic (Day 90)
  Intraclass correlation coefficient (ICC) to assess the reproducibility between the Mobile Cognition Test performed at hospital and at home
  * At Day 0 and Day 1
  * At Day 89 and Day 90
  Higher is the score, better is the outcome.
Correlation of the reproductibility of MSCopilot Boost functional test from the hospital to home. | During the first in-clinic visit (Day 0), the first at-home visit (Day 1), the follow-up visit at-home (Day 89) and the follow-up visit in-clinic (Day 90)
  Intraclass correlation coefficient (ICC) to assess the reproducibility between the Mobile Vision Test performed at hospital and at home
  * At Day 0 and Day 1
  * At Day 89 and Day 90
  Higher is the number or letter stated, better is the outcome.
To evaluate the test-retest reliability of MSCopilot Boost functional test performed at home. | During the at-home follow-up visits (Day 30, Day 60, Day 120, Day 150, Day 210 and Day 240)
  Intra class correlation coefficient coefficient will be used to evaluate the reliability of the Mobile walking perimeter test (in meter) performed at home at Day 30, Day 60, Day 120, Day 150, Day 210 and Day 240.
  Higher is the distance, better is the outcome.
To evaluate the test-retest reliability of MSCopilot Boost functional test performed at home. | During the at-home follow-up visits (Day 30, Day 60, Day 120, Day 150, Day 210 and Day 240)
  Intra class correlation coefficient coefficient will be used to evaluate the reliability of the Mobile Dexterity Test (in seconds) performed at home at Day 30, Day 60, Day 120, Day 150, Day 210 and Day 240.
  Shorter is the time, better is the outcome.
To evaluate the test-retest reliability of MSCopilot Boost functional test performed at home. | During the at-home follow-up visits (Day 30, Day 60, Day 120, Day 150, Day 210 and Day 240)
  Intra class correlation coefficient coefficient will be used to evaluate the reliability of the Mobile cognition Test (score) performed at home at Day 30, Day 60, Day 120, Day 150, Day 210 and Day 240.
  Higher is the score, better is the outcome.
To evaluate the test-retest reliability of MSCopilot Boost functional tests performed at home. | During the at-home follow-up visits (Day 30, Day 60, Day 120, Day 150, Day 210 and Day 240)
  Intra class correlation coefficient coefficient will be used to evaluate the reliability of the Mobile vision test (number of letter stated) performed at home at Day 30, Day 60, Day 120, Day 150, Day 210 and Day 240.
  Higher is the number or letter stated, better is the outcome.
To evaluate the test-retest reliability of MSCopilot Boost functional tests performed at home. | During the at-home follow-up visits (Day 30, Day 60, Day 120, Day 150, Day 210 and Day 240)
  Intra class correlation coefficient coefficient will be used to evaluate the reliability of the Mobile Walking Endurance test (in meters) performed at home at Day 30, Day 60, Day 120, Day 150, Day 210 and Day 240.
  Higher is the distance, better is the outcome.
To assess the number of adverse events of using MSCopilot Boost. | Throughout the study for all visits in-clinic (Day 0, Day 90, Day 180 and Day 270) and at-home visits (Day 1, D 30, Day 60, Day 89, Day 120, Day 150, Day 210 and Day 240)
  The application's safety of use will be assessed through a descriptive analysis of adverse events and Adverse Events associated with its use. Data relative to Adverse Events will be reported on a table, numbers and percentages reported for each group, categorizing Adverse Events as mild, moderate and severe. A descriptive analysis of risk questionnaire responses in the Boost group will also be performed.
To compare the effect of MSCopilot Boost on walking compared to standard practice: -Assessed by the functional standard test performed at the hospital -Assessed at home | During the first in-clinic visit (Day 0), during the in-clinic follow-up visits (Day 90 and Day180) and the end of study visit in-clinic (Day 270)
  Comparison of mean improvement in results between the two groups:
  * For the Timed 25 Foot Walk test (in seconds)
  * Between Day 0 and Day 90
  * Between Day 0 and Day 180
  * Between Day 0 and Day 270
  * Measured by actimeter:
  * Between Day 0 and Day 90
  * Between Day 0 and Day 180
  * Between Day 0 and Day 270
  Shorter is the time, better is the outcome.
To compare the proportion of patients whose symptoms improved in both groups on Fatigue impact. | During the first in-clinic visit (Day 0), during the in-clinic follow-up visits (Day 90 and Day180) and the end of study visit in-clinic (Day 270)
  Comparison of patients considered as improved at Day 90, Day 180 and Day 270 in both groups on the Modified Fatigue Impact Scale (MFIS)
  The score ranges from 0 to 84, with a higher score indicating a worse outcome.
To compare the proportion of patients whose symptoms improved in both groups on anxiety and depression. | During the first in-clinic visit (Day 0), during the in-clinic follow-up visits (Day 90 and Day180) and the end of study visit in-clinic (Day 270)
  Comparison of patients considered as improved at Day 90, Day 180 and Day 270 in both groups on the Patient Health Questionnaire-4 (PHQ-4)
  Score ranges from 0 to 12, with higher score indicating worse outcome.
To compare the proportion of patients whose symptoms improved in both groups on Depression. | During the first in-clinic visit (Day 0), during the in-clinic follow-up visits (Day 90 and Day180) and the end of study visit in-clinic (Day 270)
  Comparison of patients considered as improved at Day 90, Day 180 and Day 270 in both groups on the Beck Depression Inventory - Fast Screen (BDI- FS).
  The score ranges from 0 to 21, with higher score indicating worse outcome.
To compare the proportion of patients whose symptoms improved in both groups on Fatigue. | During the first in-clinic visit (Day 0), during the in-clinic follow-up visits (Day 90 and Day180) and the end of study visit in-clinic (Day 270)
  Comparison of patients considered as improved at Day 90, Day 180 and Day 270 in both groups on Fatigue with visual analog scale (from daily activities impact questionnaire)
  The score ranges from 0 to 10, with higher score indicating worse outcome.
To compare the proportion of patients whose symptoms improved in both groups on Walking. | During the first in-clinic visit (Day 0), during the in-clinic follow-up visits (Day 90 and Day180) and the end of study visit in-clinic (Day 270)
  Comparison of patients considered as improved at Day 90, Day 180 and Day 270 in both groups on the Timed 25 Foot Walk test (in seconds).
  Shorter is the time, better is the outcome.
To compare the proportion of patients whose symptoms improved in both groups on Dexterity. | During the first in-clinic visit (Day 0), during the in-clinic follow-up visits (Day 90 and Day180) and the end of study visit in-clinic (Day 270)
  Comparison of patients considered as improved at Day 90, Day 180 and Day 270 in both groups on the 9 Hole Peg Test (in seconds).
  Shorter time indicating better outcome.
To compare the proportion of patients whose symptoms improved in both groups on Cognition. | During the first in-clinic visit (Day 0), during the in-clinic follow-up visits (Day 90 and Day180) and the end of study visit in-clinic (Day 270)
  Comparison of patients considered as improved at Day 90, Day 180 and Day 270 in both groups on the Symbol Digit Modalities Test.
  Higher is the score, better is the outcome.
To compare the proportion of patients whose symptoms improved in both groups on the Low-contrast Vision. | During the first in-clinic visit (Day 0), during the in-clinic follow-up visits (Day 90 and Day180) and the end of study visit in-clinic (Day 270)
  Comparison of patients considered as improved at Day 90, Day 180 and Day 270 in both groups on the Sloan Low Contrast Letter Acuity Test (number stated).
  Higher is the number or letter stated, better is the outcome.
To compare the effect of MSCopilot Boost on quality of life compared to standard practice. | During the first in-clinic visit (Day 0), during the in-clinic follow-up visits (Day 90 and Day180) and the end of study visit in-clinic (Day 270)
  Comparison of mean improvement in EQ5D-5L results between the two groups:
  * Between Day 0 and Day 90
  * Between Day 0 and Day 180
  * Between Day 0 and Day 270
  The scale ranges from 0 to 100, with higher score means better outcome.
To compare the effect of MSCopilot Boost on the mean overall physical activity compared to standard practice. | During the first in-clinic visit (Day 0), during the in-clinic follow-up visits (Day 90 and Day180) and the end of study visit in-clinic (Day 270)
  Comparison of the evolution of the mean overall physical activity in Metabolic Equivalent of Task (MET) measured by actimeter between the two groups:
  * Between Day 0 and Day 90
  * Between Day 0 and Day 180
  * Between Day 0 and Day 270
To evaluate the satisfaction and user experience of both patients and healthcare professionals regarding MSCopilot Boost. | During at-home follow-up visit (Day 30) and in-clinic visits (Day 180 and Day 270)
  Descriptive analysis of responses collected from satisfaction and user experience questionnaires in the Boost group and from healthcare professionals.
  Each answer propose a scale from 1 to 5 or 1 to 10. Higher score means better outcome.
To assess the clinical benefit of MSCopilot Boost reported by patients and healthcare professionals. | During the end of study visit in-clinic (Day 270)
  Descriptive analysis of collected responses from clinical benefit questionnaires in Boost group and from healthcare professionals.
  Each answer propose a scale form 1 to 10 with higher score means better outcome.
To assess the organizational impact of MSCopilot Boost as reported by healthcare professionals. | During the end of study visit in-clinic (Day 270)
  Descriptive analysis of collected responses from organizational impact questionnaire administered to healthcare professionals.
  Each answer propose 5 levels of intensity from totally disagree to totally agree.
To assess user compliance with MSCopilot Boost throughout the follow-up period. | Throughout the study for all visits in-clinic (Day 0, Day 90, Day 180 and Day 270) and at-home visits (Day 1, D 30, Day 60, Day 89, Day 120, Day 150, Day 210 and Day 240)
  Number of completed evaluations per quarter compared to the theoretical maximum completion expected over time in the Boost group:
  * Functional tests
  * Fatigue evaluation questionnaires
  * Fatigue management program (tips and physical activity program)

OTHER OUTCOMES:
To evaluate the link between MSCopilot Boost use compliance and fatigue improvement. | Throughout the study for all visits in-clinic (Day 0, Day 90, Day 180 and Day 270) and at-home visits (Day 1, D 30, Day 60, Day 89, Day 120, Day 150, Day 210 and Day 240)
  Correlation coefficient between MSCopilot Boost use compliance and Modified Fatigue Impact Scale score and comparison of the mean compliance pourcentage between patients who experienced a clinically significant improvement in fatigue and those who did not.
To assess the relationship between self-reported and objectively measured physical activity. | Throughout the study from Day 0 to Day 270
  Correlation coefficient between self-reported physical activity in MSCopilot Boost and objectively measured physical activity by actimeter in the Boost group.
To explore the factors that might influence the effect of MSCopilot Boost on fatigue and its impact. | During the first in-clinic visit (Day 0) and the end of study visit in-clinic (Day 270)
  Evaluation of the interaction terms between the Boost patient group versus the control patient group and covariates (socio-demographic characteristics, depression, compliance, physical activity, etc…) in a multivariate regression model with response variables:
  * The Modified Fatigue Impact Scale score
  * Fatigue with Visual analog scale score (from daily activities impact questionnaire)
To assess the changes in sleep patterns and areas of life impacted by fatigue, as measured with MSCopilot Boost at home. | Throughout the study for all visits in-clinic (Day 0, Day 90, Day 180 and Day 270) and at-home visits (D 30, Day 60, Day 120, Day 150, Day 210 and Day 240)
  Descriptive analysis of responses collected from sleep and daily activities questionnaires in the Boost group.
  Visual Analog Scale ranges from 0 (not impacted) to 10 (very impacted), with a higher score indicating a worse outcome.
To assess the evolution of overall physical activity reported by patients. | Throughout the study from Day 0 to Day 270
  Measure of the average self-reported overall physical activity in MSCopilot Boost application each week between Day 0 and Day 270 by the Boost group.
To explore the correlation between overall physical activity and the change in : -Fatigue impact -Fatigue | During the first in-clinic visit (Day 0) and the end of study visit in-clinic (Day 270)
  Correlation coefficient assessed between the Modified Fatigue Impact Scale and physical activity (Self-reported and measured by actimeter) with the scores on the fatigue reported with a visual analog scale (from daily activities impact questionnaire) and physical activity (Self-reported and measured by actimeter).
  Visual analog scale ranges from 0 to 10. Higher score means better outcome.
Calculation of cost-effectiveness in reducing fatigue at 1, 3, 6 and 9 months using MSCopilot Boost as an intervention, compared to standard care. | During the first in-clinic visit (Day 0), during the in-clinic follow-up visits (Day 90 and Day180) and the end of study visit in-clinic (Day 270)
  Average cost mean (estimated by the number and type of hospital admissions and unscheduled medical visits) between the two groups, adjusted for the difference of quality of life between the two groups.
To assess the impact of MSCopilot Boost on work-related factors (duration without working, absenteeism from work, return-to-work time, presenteeism) at 3, 6 and 9 months, compared to baseline (Day 0), in both groups. | During the first in-clinic visit (Day 0), during the in-clinic follow-up visits (Day 90 and Day180) and the end of study visit in-clinic (Day 270)
  Mean duration without working, average number of absenteeism days, average return-to-work time, and presenteeism duration within the past 6 months will be calculated at Day 0, Day 90, Day 180 and Day 270.
To evaluate behavioral changes in terms of physical activity and energy management. | During the first in-clinic visit (Day 0), during the follow-up at-home visit (Day 30), during the follow-up in-clinic visits (Day 90 and Day180) and the end of study visit in-clinic (Day 270)
  Comparison of physical activity volume and energy-saving management routines at Day 0, Day 30, Day 90, Day 180 and Day 270 in both groups.